CLINICAL TRIAL: NCT02252211
Title: A Phase I Safety and Bioimaging Trial of DS-8895a in Patients With Advanced or Metastatic EphA2 Positive Cancers
Brief Title: Safety and Bioimaging Trial of DS-8895a in Patients With Advanced EphA2 Positive Cancers
Acronym: LUD2014-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry); Austin Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2014-002
Record Dates: First submitted 2014-09-22; First posted 2014-09-30 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Malignant Solid Tumor; Metastatic EphA2 Positive Cancer
Keywords: EphA2 positive cancer; DS-8895a monoclonal antibody

STUDY DESIGN:
Intervention Model Description: Patients were enrolled in sequential cohorts following a 3+3 dose-escalation scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DS-8895a (Experimental): Patients received infusions with DS-8895a on Days 1, 8, 22, and 36. Infusions on Days 1 and 36 were trace labelled with ^89Zr (^89Zr-Df-DS-8895a). The Day 1 dose was 0.2 mg/kg, followed by subsequent doses calculated based on individual patient body weight and dosing cohort assignment.
  Interventions: Drug: DS-8895a 1 mg/kg; Drug: DS-8895a 3 mg/kg; Drug: DS-8895a 10 mg/kg

INTERVENTIONS:
Drug: DS-8895a 1 mg/kg — Patients received infusions with ^89Zr-Df-DS-8895a at a dose of 0.2 mg/kg on Day 1, DS-8895a at a dose of 1 mg/kg on Days 8 and 22, and ^89Zr-Df-DS-8895a at a dose of 1 mg/kg on Day 36. Patients who responded or had stable disease per RECIST version 1.1 at the Day 50 restaging may have continued to receive biweekly treatment with DS-8895a until disease progression.
Drug: DS-8895a 3 mg/kg — Patients received infusions with ^89Zr-Df-DS-8895a at a dose of 0.2 mg/kg on Day 1, DS-8895a at a dose of 3 mg/kg on Days 8 and 22, and ^89Zr-Df-DS-8895a at a dose of 3 mg/kg on Day 36. Patients who responded or had stable disease per RECIST version 1.1 at the Day 50 restaging may have continued to receive biweekly treatment with DS-8895a until disease progression.
Drug: DS-8895a 10 mg/kg — Patients were to receive infusions with ^89Zr-Df-DS-8895a at a dose of 0.2 mg/kg on Day 1, DS-8895a at a dose of 10 mg/kg on Days 8 and 22, and ^89Zr-Df-DS-8895a at a dose of 10 mg/kg on Day 36. Patients who responded or had stable disease per RECIST version 1.1 at the Day 50 restaging may have continued to receive biweekly treatment with DS-8895a until disease progression.

SUMMARY:
This was a Phase 1, dose-escalation, non-randomized, open-label, single-center study of DS-8895a in patients with advanced or metastatic Ephrin type-A receptor 2 (EphA2)-positive cancers. The primary study objective was to determine the safety of DS-8895a, with secondary objectives of determining the biodistribution, tumor uptake (bioimaging), pharmacokinetics (PK), antitumor and pharmacodynamic response, and correlations between pharmacodynamics and clinical outcomes, as appropriate.

DETAILED DESCRIPTION:
Patients received an initial ^89Zr trace-labelled infusion of DS-8895a on Day 1, followed by safety assessments, positron emission tomography (PET) imaging, and PK sampling over a 1-week period. DS-8895a was infused again on Days 8, 22, and 36. The Day 36 infusion of DS-8895a was also trace labelled with ^89Zr, with subsequent PET imaging and PK sampling. Four dose levels (1, 3, 10 and 20 mg/kg) were to be evaluated, with 3 to 6 patients entered at each dose level. Patients who responded or had stable disease per the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 at the Day 50 restaging may have continued to receive biweekly treatment with DS-8895a until disease progression, with restaging performed by computed tomography (CT) scans every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced or metastatic EphA2 positive cancer (based on immunohistochemistry of archived or fresh tumor tissue).
2. Malignant tumor that was refractory to standard treatment.
3. At least one reference tumor > 1 cm in size for assessment of tumor uptake of ^89Zr-Df-DS-8895a.
4. Expected survival of at least 3 months.
5. Eastern Cooperative Oncology Group performance status ≤ 1.
6. Within the last week prior to the first study drug administration, laboratory parameters for vital functions were to be in the normal range. Out-of-range values that were not clinically significant were permitted, except that the following parameters were to be in the specified ranges:

   * Neutrophil count ≥ 1.5 x 10^9/L
   * Platelet count ≥ 90 x 10^9/L
   * International normalized ratio ≤ 1.5
   * Serum aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x the upper limit of normal (ULN); ≤ 5 x ULN if liver metastases
   * Serum bilirubin ≤ 1.5 x ULN
7. Calculated creatinine clearance ≥ 55 mL/min.
8. Age ≥ 18 years.
9. Able and willing to give valid written informed consent.

Exclusion Criteria:

1. Active central nervous system metastases. Definitively treated metastases were allowed if stable for 6 weeks off therapy.
2. Known immunodeficiency or human immunodeficiency virus positivity.
3. Serious illnesses, e.g., serious infections requiring antibiotics, bleeding disorders, or any condition that in the opinion of the Investigator would have interfered with the ability of the patient to fulfill the study requirements.
4. Other malignancy, apart from non-melanoma skin cancer, within 3 years prior to the first study drug administration that in the opinion of the investigator had > 10% risk of relapse within 12 months.
5. Significant allergic reaction to prior antibody infusions.
6. Chemotherapy, radiotherapy, or investigational agent within 4 weeks prior to the first study drug administration.
7. Regular corticosteroid, non-steroidal anti-inflammatory drug (other than paracetamol or low-dose aspirin) or other immunosuppressive treatment within 3 weeks prior to the first study drug administration (intermittent dosing permitted if less than 4 doses within a 3-day period).
8. Mental impairment that could have compromised the ability to give informed consent and comply with the requirements of the study.
9. Lack of availability for clinical follow-up assessments.
10. Pregnancy or breastfeeding.
11. Women of childbearing potential: Refusal or inability to use effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2016-09-08 (Actual); Study Completion 2016-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Scott, MD, Principal Investigator — Austin Health, Melbourne, Australia; Hui Gan, MD, PhD, Principal Investigator — Austin Health, Melbourne, Australia
Locations (1):
- Austin Health, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gan HK, Parakh S, Lee FT, Tebbutt NC, Ameratunga M, Lee ST, O'Keefe GJ, Gong SJ, Vanrenen C, Caine J, Giovannetti M, Murone C, Scott FE, Guo N, Burvenich IJG, Paine C, Macri MJ, Kotsuma M, Senaldi G, Venhaus R, Scott AM. A phase 1 safety and bioimaging trial of antibody DS-8895a against EphA2 in patients with advanced or metastatic EphA2 positive cancers. Invest New Drugs. 2022 Aug;40(4):747-755. doi: 10.1007/s10637-022-01237-3. Epub 2022 Apr 11. PMID 35404015

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg | DS-8895a 10 mg/kg
Started | 5 | 3 | 1
Received Dose 1 (Day 1) | 4 | 3 | 0
Received Dose 2 (Day 8) | 4 | 3 | 0
Received Dose 3 (Day 22) | 3 | 3 | 0
Received Dose 4 (Day 36) | 1 | 1 | 0
Received Further Doses (Through Dose 24) | 1 | 0 | 0
Completed (Completed the study as planned per protocol) | 0 | 0 | 0
Not Completed | 5 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Progressive disease | 3 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Serious Adverse Event During Screening | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set comprised all patients who received at least 1 infusion of DS-8895a.
Groups:
- Total: Total of all reporting groups
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (7.4) | 64.0 (15.1) | 65.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 4 | 3 | 7
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.4 (4.2) | 28.1 (6.4) | 26.0 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-emergent Adverse Events
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0. Treatment-emergent adverse events (TEAEs) were reported based on clinical laboratory tests, physical examinations, and vital signs from pre-treatment through the study period.
Time Frame: Continuously for up to 58 weeks
Population: The Safety Analysis Set comprised all patients who received at least 1 infusion of DS-8895a.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 4 | 3
Participants
  Any TEAE | 4 | 3
  Maximum grade 1 TEAE | 0 | 1
  Maximum grade 2 TEAE | 4 | 1
  Maximum grade 5 TEAE | 0 | 1
  Treatment-related TEAE | 0 | 0
  Treatment-emergent Serious Adverse Event | 0 | 1
  TEAE leading to study withdrawal | 0 | 1

2. Secondary Outcome: Number of Patients With Tumor Uptake of ^89Zr-Df-DS-8895a
Description: The biodistribution and tumor uptake of ^89Zr-Df-DS-8895a was determined based on qualitative analysis of whole body positron emission tomography (PET)/computed tomography (CT) images. PET imaging was performed following the ^89Zr-Df-DS-8895a infusions on Day 1 (Days 1, 4/5, and 7/8) and Day 36 (Days 36, 39/40 and 42/43). Qualitative parameters assessed included tumor uptake of reference lesions (scored on a 0-3 point scale: none, low, med, high). The reference lesions were initially identified on fluorodeoxyglucose (FDG) PET scans with a score of 3 for [18F]-fluorodeoxyglucose uptake. The summary table presents the maximum reference lesion ^89Zr-Df-DS-8895a uptake score reported for individual patients.
Time Frame: Up to Day 43
Population: The Safety Analysis Set comprised all patients who received at least 1 infusion of DS-8895a.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 4 | 3
Participants
  Maximum Lesion Uptake Score 0 (No Uptake) | 0 | 0
  Maximum Lesion Uptake Score 1 | 4 | 2
  Maximum Lesion Uptake Score 2 | 0 | 0
  Maximum Lesion Uptake Score 3 | 0 | 1

3. Secondary Outcome: Number of Patients With Best Overall Tumor Response
Description: Tumor responses were evaluated using computed tomography and categorized according to the Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1) at Screening (up to 21 days before the first dose of study drug), on Day 50, and approximately every 6 weeks thereafter for patients who received continued study dosing. Per RECIST, target lesions are categorized as follows: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Up to 58 weeks
Population: The Evaluable Analysis Set comprised all patients who received at least 1 infusion of DS-8895a and completed all study procedures up to Day 50.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 1 | 1
Participants
  Stable disease | 1 | 0
  Progressive disease | 0 | 1

4. Secondary Outcome: Mean Area Under the Serum Concentration Curve of ^89Zr-Df-DS-8895a Following the First Infusion
Description: The pharmacokinetics (PK) of ^89Zr-Df-DS-8895a were calculated based on data from gamma counting of serum samples. Serum samples for gamma counting were drawn on Day 1 (pre-infusion and 5 minutes, 1, 2, and 4 hours post-infusion), Day 2 (24 hours post-infusion), Day 4/5 (anytime), Day 36 (pre-infusion, and 5 minutes, 1, 2, and 4 hours post infusion), Day 37 (24 hours post-infusion), Day 39/40 (anytime), Day 42/43 (anytime), and Day 50 (anytime). For Cycle 2 onward, blood samples for PK were taken at pre- and 0 to 30 minutes post-infusion on Days 1, 15, and 29.
Time Frame: Cycle 1 Day 1 (pre-infusion and 5 minutes, 1, 2, and 4 hours post-infusion)
Population: The PK Analysis Set comprised all patients who received at least 1 infusion of DS-8895a and had evaluable PK samples for a given analysis.
Measure: Mean (Standard Deviation); unit: hr*μg/mL
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 4 | 3
hr*μg/mL | 349.0 (24.6) | 486.5 (169.7)

5. Secondary Outcome: Mean Volume of Distribution at Steady State of ^89Zr-Df-DS-8895a Following the First Infusion
Description: The PK of ^89Zr-Df-DS-8895a was calculated based on data from gamma counting of serum samples. Serum samples for gamma counting were drawn on Day 1 (pre-infusion and 5 minutes, 1, 2, and 4 hours post-infusion), Day 2 (24 hours post-infusion), Day 4/5 (anytime), Day 36 (pre-infusion, and 5 minutes, 1, 2, and 4 hours post infusion), Day 37 (24 hours post-infusion), Day 39/40 (anytime), Day 42/43 (anytime), and Day 50 (anytime). For Cycle 2 onward, blood samples for PK were taken at pre- and 0 to 30 minutes post-infusion on Days 1, 15, and 29.
Time Frame: Cycle 1 Day 1 (pre-infusion and 5 minutes, 1, 2, and 4 hours post-infusion)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 4 | 3
mL/kg | 64.3 (7.4) | 51.3 (16.8)

6. Secondary Outcome: Mean Total Serum Clearance of ^89Zr-Df-DS-8895a Following the First Infusion
Description: as for outcome 5
Time Frame: Cycle 1 Day 1 (pre-infusion and 5 minutes, 1, 2, and 4 hours post-infusion)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 4 | 3
mL/hr/kg | 0.6 (0.0) | 0.5 (0.2)

7. Secondary Outcome: Mean Maximum Serum Concentration of ^89Zr-Df-DS-8895a Following the First Infusion
Description: as for outcome 5
Time Frame: Cycle 1 Day 1 (pre-infusion and 5 minutes, 1, 2, and 4 hours post-infusion)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 4 | 3
µg/mL | 3.1 (0.4) | 4.2 (1.2)

8. Secondary Outcome: Mean Elimination Half-life of ^89Zr-Df-DS-8895a Following the First Infusion
Description: as for outcome 5
Time Frame: Cycle 1 Day 1 (pre-infusion and 5 minutes, 1, 2, and 4 hours post-infusion)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 4 | 3
hr | 77.4 (5.1) | 79.9 (8.3)

9. Secondary Outcome: Mean Area Under the Serum Concentration Curve of DS-8895a Following the First Infusion
Description: The PK of DS-8895a was calculated based on data from enzyme-linked immunosorbent assay (ELISA) of serum samples. Serum samples for ELISA were drawn at the same times as for gamma counting with the addition of Day 8 (pre- and 0 to 30 minutes post-infusion), Day 9 (anytime), and Day 22 (pre- and 0 to 30 minutes post-infusion). For Cycle 2 onward, blood samples for PK were taken at pre- and 0 to 30 minutes post-infusion on Days 1, 15, and 29.
Time Frame: Cycle 1 Day 1 (pre-infusion and 5 minutes, 1, 2, and 4 hours post-infusion)
Population: The PK Analysis Set comprised all patients who received at least 1 infusion of DS-8895a and had evaluable PK samples for a given analysis. One patient in the 1 mg/kg cohort did not have adequate samples to calculate PK parameters for this analysis.
Measure: Mean (Standard Deviation); unit: hr*μg/mL
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 3 | 3
hr*μg/mL | 255.2 (14.5) | 391.0 (190.0)

10. Secondary Outcome: Mean Volume of Distribution at Steady State of DS-8895a Following the First Infusion
Description: as for outcome 9
Time Frame: Cycle 1 Day 1 (pre-infusion and 5 minutes, 1, 2, and 4 hours post-infusion)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 3 | 3
mL/kg | 51.8 (8.7) | 42.1 (11.7)

11. Secondary Outcome: Mean Total Serum Clearance of DS-8895a Following the First Infusion
Description: as for outcome 9
Time Frame: Cycle 1 Day 1 (pre-infusion and 5 minutes, 1, 2, and 4 hours post-infusion)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 3 | 3
mL/hr/kg | 0.6 (0.1) | 0.5 (0.3)

12. Secondary Outcome: Mean Maximum Serum Concentration of DS-8895a Following the First Infusion
Description: as for outcome 9
Time Frame: Cycle 1 Day 1 (pre-infusion and 5 minutes, 1, 2, and 4 hours post-infusion)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 3 | 3
µg/mL | 3.0 (0.3) | 4.0 (1.2)

13. Secondary Outcome: Mean Elimination Half-life of DS-8895a Following the First Infusion
Description: as for outcome 9
Time Frame: Cycle 1 Day 1 (pre-infusion and 5 minutes, 1, 2, and 4 hours post-infusion)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 3 | 3
hr | 59.3 (9.2) | 65.3 (20.6)

14. Secondary Outcome: Number of Patients With Pharmacodynamic (Metabolic) Response
Description: The pharmacodynamic (metabolic) response of DS-8895a was assessed by ^18F-FDG PET at Screening, Day 29, and Day 50. Tumor metabolism response was evaluated as the difference in standardized uptake values between the pre- and post-treatment FDG PET scans. The measurement of [18F]-FDG uptake for tumor metabolic response monitoring was performed according to the European Organization for Research and Treatment of Cancer (EORTC) PET response criteria (Young et al. Eur J Cancer 1999;35:1773-82).
Time Frame: Day 29 and Day 50
Population: The Safety Analysis Set comprised all patients who received at least 1 infusion of DS-8895a.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 4 | 3
Participants
  Stable Disease at Days 29 and 50 | 1 | 0
  Stable Disease at Day 29, Progression at Day 50 | 0 | 1
  Progressive Disease at Day 29 | 3 | 2

15. Secondary Outcome: Number of Patients With Human Anti-Human Antibody Positivity
Description: Blood samples to detect human anti-human antibody (HAHA) formation were collected on Days 1 (pre-infusion [within 7 days of Day 1 dose] and post-infusion), 8, 22, 36 (pre-infusion), and 50 (anytime). For Cycle 2 onward, HAHA samples were collected on Day 1 (pre-infusion) and at the end of the study (anytime). HAHA samples were analyzed using ELISA and were categorized as either positive or negative for a HAHA response. HAHA positivity indicates that a patient has developed an antibody response.
Time Frame: Up to 43 Weeks
Population: The Safety Analysis Set comprised all patients who received at least 1 infusion of DS-8895a.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg
Number analyzed (Participants) | 4 | 3
Participants
  Positive HAHA Results (Single Sample) | 1 | 1
  Negative HAHA Results at all Time Points | 3 | 2

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs). The AE reporting period for this study was up to 58 weeks.
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 4.0), seriousness, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per patient at the maximum reported grade.
Groups:
- DS-8895a 1 mg/kg: Patients received infusions with ^89Zr-Df-DS-8895a at a dose of 0.2 mg/kg on Day 1, DS-8895a at a dose of 1 mg/kg on Days 8 and 22, and ^89Zr-Df-DS-8895a at a dose of 1 mg/kg on Day 36. Patients who responded or had stable disease per RECIST version 1.1 at the Day 50 restaging may have continued to receive biweekly treatment with DS-8895a until disease progression.
  All enrolled patients are included in AE tabulations; 1 patient was enrolled but discontinued due to SAEs prior to receiving study treatment.
- DS-8895a 3 mg/kg: Patients received infusions with ^89Zr-Df-DS-8895a at a dose of 0.2 mg/kg on Day 1, DS-8895a at a dose of 3 mg/kg on Days 8 and 22, and ^89Zr-Df-DS-8895a at a dose of 3 mg/kg on Day 36. Patients who responded or had stable disease per RECIST version 1.1 at the Day 50 restaging may have continued to receive biweekly treatment with DS-8895a until disease progression.
  All enrolled patients are included in AE tabulations.
- DS-8895a 10 mg/kg: Patients were to have received infusions with ^89Zr-Df-DS-8895a at a dose of 0.2 mg/kg on Day 1, DS-8895a at a dose of 10 mg/kg on Days 8 and 22, and ^89Zr-Df-DS-8895a at a dose of 10 mg/kg on Day 36. Patients who responded or had stable disease per RECIST version 1.1 at the Day 50 restaging may have continued to receive biweekly treatment with DS-8895a until disease progression.
  All enrolled patients are included in AE tabulations; 1 patient was enrolled but discontinued due to an SAE prior to receiving study treatment.
Arm/Group | DS-8895a 1 mg/kg | DS-8895a 3 mg/kg | DS-8895a 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/5 | 1/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/3 | 1/1
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-8895a 1 mg/kg (N=5) | DS-8895a 3 mg/kg (N=3) | DS-8895a 10 mg/kg (N=1)
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 — Grade 3
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — Grade 5
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 — Grade 3, not treatment emergent
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 — Grade 3, not treatment emergent
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 — Grade 5, not treatment emergent
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — Grade 3, not treatment emergent
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-8895a 1 mg/kg (N=5) | DS-8895a 3 mg/kg (N=3) | DS-8895a 10 mg/kg (N=1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0
Rectal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Crepitations (General disorders) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less